CLINICAL TRIAL: NCT00453466
Title: Group Empowerment of Battered Women as a Tool for Violence Prevention
Acronym: EBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CWHSP-03-2001
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2007-03

CONDITIONS: Domestic Violence
Keywords: women experiencing domestic violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: EBW group intervention to empower battered women

SUMMARY:
Intimate partner violence against women is a significant global health problem. This study was designed to test the hypothesis that a group intervention based on empowerment theory of Paolo Freire would be effective as a means to reduce the extent and prevent violence among women whose partners were violent toward them.

DETAILED DESCRIPTION:
A randomized controlled trial (N=141) with two control groups (one individual psychotherapeutic treatment and the other a usual care group treatment) was conducted in a violence treatment center in the South of Israel The treatment protocol designed to empower battered women (EBW) was conducted with 12 groups over a period of two years. Assessments were made before, immediately following and at an 8 month follow up following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women living in the south, who had approached the center for help as battered women
* Could fill out forms in Hebrew
* Aged 20 and above

Exclusion Criteria:

* Age younger than 20
* Not able to fill out forms in Hebrew
* Not living in the southern district of Israel

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Conflict tactics scale, Posttraumatic stress scale for
family violence

CONTACTS AND LOCATIONS:
Overall Officials: Julie G Cwikel, Ph.D., Study Director — Ben-Gurion University of the Negev